# Hydroxyurea Adherence for Personal Best in Sickle Cell Disease (HABIT): Efficacy Trial

NCT03462511

July 14, 2020

#### SPECIFIC AIMS

Sickle cell disease (SCD) is a major chronic illness affecting approximately 100,000 Americans of African descent, including Caribbean Latinos and other underserved ethnicities. An inherited blood disease, SCD is characterized by fatigue, painful crises, organ damage, reduced quality of life (QOL) and high health care costs and shortened lifespan. The sole FDA-approved drug for SCD therapy is hydroxyurea (HU); its use is recommended as standard practice. HU markedly reduces symptoms, morbidity and mortality, improves QOL, decreases health care cost, and may protect against cumulative disease burden. HU induces a dose-dependent increase in fetal hemoglobin (HbF), an effect that is largely responsible for its impact. Despite benefits of HU, adherence in adolescents and young adults is often poor. Despite benefits of HU, adherence in adolescents and young adults is often poor. Despite benefit, Des

The scientific premise and experience for the proposed study is based on our 2-site randomized feasibility trial of "HABIT" (R21NR013745), a 6-month intervention delivered by community health workers (CHWs), augmented by tailored text messages sent to subjects.<sup>31</sup> A multi-ethnic sample of 28 youth-parent dyads (youth ages 10-18 years) participated in this study. Eligible youth had ≥20% decrease from maximum HU-induced HbF levels, "Personal Best." The intervention was both feasible and acceptable, and sufficiently effective on our primary outcome of medication adherence - operationalized by two objective measures. Building on these promising results and partnering with three additional clinical sites, we propose a larger 5 site randomized controlled trial of 104 youth-parent dyads to test the efficacy of the HABIT intervention.

### Study aims are to:

**Aim 1**: Improve daily HU adherence, the primary outcome operationalized two ways: biomarker (approach or exceed a historical Personal best HbF) and pharmacy refill (proportion of days covered). <u>Hypothesis 1</u>: Compared to the control group, youth-parent dyads randomized to the intervention will improve medication adherence at 6 months, with sustained improvement at 12 months.

**Aim 2**: Improve quality of life and self-management responsibility measured by three *secondary outcomes*: generic and disease-specific QOL and parent/youth concordance regarding delegation of self-management responsibility. *Hypothesis 2*: Compared to the control group, dyads randomized to the intervention will report improved quality of life and self-management responsibility concordance at 6 months, with sustained improvement at 12 months.

**Aim 3**: Improve health status measured by two secondary outcomes: acute hospital use (12 month hospital length of stay, admissions and emergency room visits) and self-reported disease symptoms (fatigue, pain interference and intensity). <u>Hypothesis 3.1</u>: Compared to the control group, youth-parent dyads randomized to the intervention group will demonstrate decreased acute hospital use at 6 months, with sustained improvement at 12 months. <u>Hypothesis 3.2</u>: Compared to the control group, dyads randomized to the intervention group will report decreased disease symptoms at 6 months, with sustained improvement at 12 months.

**Aim 4**: Qualitatively describe impact and sustainability of the intervention on developing a daily medication HU habit from the perspectives of the community health workers (CHWs) and youth-parent-dyads using focus group and individual interviews (*exploratory aim*).

**Impact:** Adherence to daily medications is a challenge for most youth with chronic health conditions and poor adherence is common.<sup>24</sup> Identifying successful ways to improve adherence to HU through developmentally appropriate self-management not only has the potential to improve the health of youth with SCD, the intervention may be transferable to underserved youth with other chronic conditions. Further, this research is consistent with NINR's strategic theme of "Self-Management: Improving Quality of Life for Individuals with Chronic Illness,"<sup>32</sup> as well as the U.S. Healthy People 2020 goals of optimizing health across the lifespan and reducing health disparities<sup>33</sup> for SCD and other conditions.

#### **RESEARCH STRATEGY**

- **A. SIGNIFICANCE** This proposal directly responds to **PA-14-029**, "Chronic Condition Self-Management in Children and Adolescents. The proposed multi-site randomized intervention trial is the next logical step from our successful feasibility trial (R21NR013745). The trial proposed here will test a replicable and scalable model for self-managing HU adherence in SCD to decrease disease morbidity and improve QOL. It could also be applied to other chronic conditions affecting underserved youth to address health disparities. Specifically:
- 1. Poor medication adherence is a widespread challenge to optimizing health outcomes in chronic disease, <sup>34</sup> rendering treatments less beneficial or even ineffective. Adherence problems are especially pronounced in underserved communities, <sup>29,30</sup> adding to existing health disparities, increased health cost expenditures <sup>34,35</sup> and decreased QOL <sup>10,36</sup> This problem is common among youth with chronic illness, especially those with social, economic, linguistic and cultural barriers. <sup>16-18,20</sup> Mismatches between providers and communities served are known risk factors for reduced adherence. <sup>20,37,38</sup> Barriers to adherence include incomplete understanding of disease and benefits to medication use, <sup>11,19,39</sup> access to medication <sup>22</sup> and poor family adaptation to chronic illness. <sup>40</sup> Adolescents with chronic medical conditions have especially high rates of poor adherence, <sup>24,26,41</sup> especially those from under-resourced communities. <sup>41</sup> Moreover, problems with self-management during adolescence interferes with successful transition to young adulthood. <sup>40,42</sup>
- **2. SCD** is a major chronic multi-organ illness, affecting approximately 100,000 African American, Hispanic and other traditionally underserved communities in the U.S. <sup>1,7,43</sup> SCD frequently affects underserved groups in the U.S.: 1:365 of African-American births and 1:16,300 of Hispanic-American births. <sup>1</sup> SCD is associated with high medical expenditures, <sup>44</sup> early mortality, poor QOL and low rates of high school completion. <sup>4</sup> Reflecting the importance of SCD to population health and reducing health disparities the federal Healthy People 2020 (HP 2020) program of goals for national health-promotion and disease prevention includes target goals for SCD. <sup>45</sup>
- **3. Youth and young adults with SCD derive considerable health benefit from HU treatment,** 8,9,46 **but poor adherence common,** 10-14,39 often reflecting poor self-management. HU benefits include reduced symptoms, 7,47 health care expenditures and improved health QOL for the common sickle subtypes (HbSS and HbS-B0 thalassemia). Increased well-being often begins within the first months of HU, along with increased HbF levels. Optimum therapeutic effect is reached at maximum HbF response, which we refer to as "Personal best HbF levels". Rarely is HU therapy ineffective in childhood, and is usually attributable to poor adherence. Young adults with SCD utilize health care at the highest levels of all age groups, including hospitalization and re-admission, and here high rates of poor adherence. Adult HU use is associated with improved outcomes and longevity, 11,52 In total, these findings demonstrate the impact of HU *across the lifespan*, underscoring the imperative of establishing self-management of HU during childhood and adolescence. Consistent with NINR's strategic theme of "Self-Management Improving Quality of Life for Individuals with Chronic Illness," HP 2020 public health goals for SCD include the increased use of disease-modifying therapies, of which HU is the most widely available effective treatment.
- **4.** If demonstrated as efficacious, our HABIT intervention could be adapted to address poor medication adherence across other chronic pediatric conditions in underserved communities. Our approach built upon Columbia's local pediatric asthma study for underserved communities in Washington Heights and Harlem. <sup>53</sup> CHW-based approaches are recommended to improve treatment outcomes for chronic pediatric conditions in underserved communities, <sup>54</sup> and need successful models for implementation.
- **B. INNOVATION**. To develop a self-managed adherence habit<sup>23</sup> for HU for youth with SCD, the proposed multi-site randomized HABIT trial will continue to employ several innovative aspects:
- **1. Individualized Personal Best HbF target**. No standard previously existed to assess HU adherence<sup>9,11,13,39,55</sup> We have used and validated the highest historical HU-induced HbF as an innovative minimum target for an individualized Personal Best self-management goal.<sup>15,31</sup> Long-term pediatric clinical HU trials demonstrated stable HbF levels over time.<sup>56-58</sup> The personalized biomarker of Personal best HbF adds to other adherence measures employed and serves as a customized motivational aid. In the HABIT feasibility trial, coaching by CHWs on the historical Personal best HbF helped create a concrete attainable goal and was useful and acceptable to youth-parent dyad participants. We validated the utility of Personal best as a biomarker for tracking adherence in a retrospective sample of 75 youth on HU therapy<sup>15</sup> (see **Preliminary studies C2**)
- **2.** Focus on underserved parent-youth dyads and developmentally appropriate delegation of responsibility for adherence. Chronic disease management often deteriorates during adolescence as youth assume greater self-management responsibility. Shared responsibility in youth-parent partnerships for self-management supports adolescents by a gradual transition to self-management. To our knowledge,

the HABIT trial is the only CHW intervention to engage youth-parent dyads.

**3.** Community Health Worker (CHW) support augmented by tailored text messaging. Our approach combines two successful research strategies for a novel multi-component approach for improved cue-based medication adherence. Culturally aligned CHWs are an accepted mode of by community-based support for improving health in underserved communities. <sup>53,66-68</sup> CHWs share responsibility for patient education, support and social services with clinical staff, and have been successful in engaging and sustaining adherence among adolescents. CHWs are highly effective at promoting adherence to chronic disease management regimens through regular, structured interactions. <sup>53</sup> Currently, CHWs are being tested a multi-state, federally funded program to improve access to care for adults with SCD (LOS **Banks**). In the HABIT feasibility trial, CHWs established a trusting relationship with families and focused on helping the youth-parent dyad work together to address their particular barriers to medication adherence.

Texting health messages is effective for professional-to-parent short-term reminders, <sup>69</sup> and are widely acceptable and effective for parents and adolescents. <sup>69,70</sup> Text-based reminders to improve adherence in chronic pediatric illnesses may improve a biomarker but have not documented changes in health status or sustainability. <sup>71</sup> Other types of electronic communication were less popular in our community for connecting youth and their parents. <sup>72</sup> During the feasibility study, HABIT dyads worked collaboratively with the CHWs to personalize automated, cue-based text messaging to reinforce the HU habit. This approach builds on work demonstrating the importance of tailored communication messages. <sup>70,73</sup> **To our knowledge, this combined intervention has not previously been studied for improving medication adherence**.

#### C. RESEARCH STRATEGY

- 1. Scientific Premise and Overall Strategy. Poor medication adherence is highly prevalent among children<sup>24</sup> and in adults<sup>74</sup> with chronic health conditions. Poor adherence poses considerable risk for exacerbating health burden, cost and health disparities. Rigorous multi-level tracking of treatment adherence and its impact includes health care utilization, treatment success rates, family functioning and school/work missed, bioassays and symptoms.<sup>75</sup> For SCD, widespread poor adherence for therapeutic HU for SCD has been documented by pharmacy refill databases<sup>10,13,76</sup> and by reduction from peak HbF levels,<sup>13,15</sup> the most sensitive biomarker for dose-dependent HU use. Systematic reviews and meta-analyses of randomized trials to improve adherence among youth with chronic illness support the importance of multi-modal approaches,<sup>77,78</sup> some of which include community-based support.<sup>53</sup> Trials to improve HU adherence are limited, and to date have focused on immediate outcomes rather than broader patient-reported outcomes, and have not used strategies for developing longer-term self-management<sup>71,79,80</sup> that are sensitive to socio-cultural patient and family needs. Using individualized biomarker and pharmacy data, we propose a rigorously designed and implemented multi-site randomized controlled trial to test the efficacy and sustainability of the intervention.
- **2. Preliminary Studies.** Our multidisciplinary team has complementary expertise, which ensures our ability to fulfill study goals. The studies that directly inform the scientific premise of this application are described below.
- a. Expertise of the Inter-disciplinary Research Team: The majority of the research team (Smaldone, Green, Jia, Findley, Manwani) and consultants (Matos, Stennett) collaborated on our successful HABIT 2-site feasibility trial. Bruzzese, with extensive experience in developing evidence-based asthma interventions to youth and their caregivers in school settings, 81-84 and Stockwell, nationally recognized for her work in text messaging interventions to improve pediatric vaccination, 69,70,85 bring their expertise to the research team. Our new site PIs Smith-Whitely, and Aygun are experienced in conducting clinical research trials, community based outreach, patient/family support and assessing patient-oriented outcomes. 24,86-88

**Table 1. Study Team and Relevant Expertise** Co-I = Co-investigator

| | Role | Discipline | SCD | Self-<br>mgmt | Adolesc<br>Transition | Community<br>Intervention | Technology in Health | Clinical<br>Trials | Qual.<br>Analysis |
|---|---|---|---|---|---|---|---|---|---|
| Green | Pls | Pediatric Sickle Cell | + | + | | + | + | + | |
| Smaldone | Pls | Nursing, Pediatrics | | + | + | + | + | + | + |
| Bruzzese | Co-I | Psychology | | + | + | + | | + | |
| Jia | Co-I | Biostatistics | | | | | | + | |
| Findley | Co-I | Public health | | + | | + | | + | + |
| Stockwell | Co-I | eHealth, texting | | | | | + | + | |
| Smith-<br>Whitely | Site PI | Pediatric Sickle Cell | + | | | + | | + | |
| Aygun | Site PI | Pediatric Sickle Cell | + | | | | | + | |
| Manwani | Site PI | Pediatric Sickle Cell | + | | | + | | + | |

| Matos | Consultant | CHW training | + |
|----------|------------|--------------------|---|
| Stennett | Consultant | Community services | + |

**b. HABIT feasibility trial**: This study (R21NR013745) tested the feasibility and acceptability of the 6-month intervention to improve adherence to HU therapy in a sample of youth-parent dyads and estimated effect size<sup>31</sup>. The intervention was highly structured to assure fidelity while also tailored for individual youth-parent dyad needs. During months 1- 6, CHWs had monthly face-to-face interactions at the subject's home or other location where privacy was assured. CHWs also met dyads at one clinic visit. To support relationship building, additional contact between dyad members and CHWs was maintained, as needed, by phone or text message by dyad member preference. CHWs communicated HbF results to the dyad soon after each test, discussed challenges to reducing barriers to HU adherence, and progress made to achieve Personal Best HbF. The structured assessment for each CHW visit is found in Appendix 6.

Tailored interactive text message reminders were collaboratively developed with each dyad member to support linking a daily cue to form a HU adherence behavior. This was initiated in month 3 to allow time for establishing the relationship with CHWs. Subjects lacking a mobile phone or sufficient cell phone plan were provided a simple cell phone or were compensated to upgrade plans to accommodate texts. Text messages were programmed to appear as sent by the CHW. Texts sent and received were tracked by the MIR3 texting system (Appendix 7).

Of 74 youth screened at 2 study sites, 48 met all inclusion/exclusion criteria and 28 dyads (58% acceptance) participated in the study. Subject attrition was 10.7%. Reasons for dyad attrition were incarceration, illicit drug activity (1 youth each) and burdensome study procedures (1 parent). On average, youth were 14.3±2.6 years, 43% female and 50% Hispanic. The majority of parents were single and/or separated from a spouse, had a high school education or less, and were employed full or part time. Spanish language surveys were used by 42% of parents and 25% of youth subjects. The 2:1 enrollment scheme allowed for more feedback about the HABIT intervention.

**Feasibility and acceptability**. Monthly CHW visits were feasible, although more frequent visits were not. Text messages were delivered as planned, once the logistical barrier of a blocked phone number was addressed.

The majority of parents and youth reported that they found meeting time with the CHW convenient, found the study's educational materials helpful, and learned new information about SCD and HU. Intervention subjects reported that they felt the CHWs valued their opinion, were easy to talk to about their disease, and helped the dyad to improve their collaboration in managing SCD. Subjects did not find the text messaging burdensome. The majority of parents (81.3%) and youth (75.1%) reported that linking the text message to the time of an activity made it easier to remember to take HU. When asked what they liked about working with the CHWs, a dyad stated "it seemed like family talking to everyone" (parent) and "it gave me a better mindset" (youth). Of 18 dyads who participated in the intervention, 10 (56%) required referrals made by CHWs. The most frequent referrals were for mental health services (n=5) and housing (n=5). CHWs met with nearly all of the dyads at their home; visits lasted 60-90 minutes. CHW visits consisted of conversations with both dyad members present, and dyads reported making progress in working together as a team. CHWs felt that a relationship was established with the majority (68%) of parents at the first visit, with most youth (81%) by the second visit and with all by the third visit.

Primary outcome: improved HU adherence. At baseline, decrease of ≥20% from Personal Best HbF (Personal best) was higher in the control group compared to the intervention group (-42.6±21.3 vs -18.1±23.6). Controlling for study month the intervention group progressed to Personal best by 2.3% per month during months 0 to 4 (p=0.31). Some subjects in the invention group even exceeded their Personal Best goal, likely due to previously inadequate HU adherence. We used improvement toward Personal Best HbF as the basis for the power analysis of the proposed multi-site trial. Results were similar when we measured adherence by Proportion of Days covered by medication (PDC) using pharmacy refill data. The intervention group improved PDC from 64.6% (year pre-enrollment) to 79.4% at month 6, an increase of 14.8%. In contrast, the control group had a smaller change of 6.5% (79.4% pre-enrollment to 85.9% at month 6).

Secondary outcomes: QOL and dyad concordance regarding self-management responsibility. From 0-6 months, both generic and disease specific QOL improved for intervention youth (generic  $+6.3\pm12.6$ , p=0.01; disease specific  $6.1\pm17.3$ , p=0.33) but not for controls ( $-2.4\pm9.1$ , p=0.57;  $-1.2\pm17.5$ , p=1.0). Controlling for month and group assignment, youth in the intervention group improved generic quality of life scores by 1.6 points/month during months 0 to 6 (p=0.02). From enrollment to 3 months, dyad self-management concordance improved for intervention dyads ( $+1.3\pm2.1$ , p=0.03) but not controls ( $0.2\pm1.6$ , p=0.80).

Value of booster session during the sustainability phase of proposed study. Parents (9 of 18) who participated in the intervention group during our HABIT feasibility trial were interviewed by telephone regarding their opinion of the value of an additional "booster" visit by the CHW. All felt that the extra CHW visit would be well accepted. The majority (89%) identified the 8 month visit as the best timing for the visit with the preferred location either at home (78%) or clinic (89%). All stated that weekly phone calls with CHWs would be accepted by parents but were not sure about weekly contact with youth.

c. Larger decline from Personal Best HbF is associated with higher urgent hospital use. To validate the concept of Personal best as a measure of HU adherence, we conducted a retrospective review of 75 youth ages 10-18 years with SCD prescribed HU at the two centers which participated in our HABIT feasibility trial. HbF was examined pre-HU initiation, at Personal Best (HbF at maximum HU dose), and recent assessment. Decrease from Personal best HbF of ≥20% at recent assessment was considered a marker of suboptimal HU adherence. In contrast, a decrease of <20% was considered stable. In all, 70% of youth (n=53) met criterion for

suboptimal adherence with average decrease from Personal Best HbF 40.1±17.5% significantly higher compared to 11.7±5.3% in the stable group, p<0.001). Those with greater decline from Personal Best HbF differed from those with more stable HbF in terms of longer time to achieve Personal Best (p=0.01), higher HU dose at Personal Best (p=0.02) and higher recent HU dose (p=0.03). Resource use was measured over two 1-year periods: at Personal Best HbF (6 months pre to post Personal Best) and at recent HbF assessment (6 months pre to post assessment). Comparing the periods for each group, urgent hospital visits and total hospital length of stay (LOS) (Figure 1) remained



stable at recent assessment for youth with low decline from Personal Best (hospital use -0.05; p=0.52; -0.6; p=0.48). However, both increased for youth with larger decline from Personal Best (hospital use +1.2; p=0.01; LOS +5.2, p=0.001). A sensitivity analysis, conducted using cutoffs of 25% and 15%, tested the robustness of study findings and yielded similar results. These data support Aim 3 of the proposed study.

d. Translation and linguistic validation of PedsQL SCD module. The PedsQL Sickle Cell disease module<sup>89</sup> became available to researchers in 2013. Due to its alignment with HABIT outcomes, we added it into the battery of survey instruments used in our feasibility study. The instrument was only available in English. Assisted by a PhD student at Columbia's School of Nursing, the 8-12 year and 13-18 year versions of the instrument underwent a forward and backward translation process. Twenty subjects (10 parents, 10 youth with SCD, half in each age group) participated in the final phase of validation. Each subject first completed the translated questionnaire and then participated in a cognitive interview to determine whether questionnaire directions, questions and response choices were clear, relevant, appropriate, and easily understood. The translated survey was well received and required no changes. The long term goal is to make the instrument available to researchers to allow participation of Spanish speaking youth with SCD and their parents. A report of the process of translation and a summary of the cognitive interviews was submitted to MAPI Institute.

## **Proposed HABIT Intervention Study:**

**3. Theoretical Frameworks.** The Self and Family Management Framework <sup>90</sup> guides the study design for Aims 1-3. Designed to better understand and improve self- and family self-management of chronic conditions, the framework addresses key youth and family risk and protective factors for youth and family. These factors include health status, individual and family factors, environmental context and developmental aspects. Recently updated, the revised framework highlights processes such as activation of resources to promote self-management of chronic illness and differentiates proximal from distal outcomes. In this study we examine the efficacy and sustainability of a community intervention employing CHWs (process) on proximal (adherence behaviors and symptom management) and distal (quality of life, self-management responsibility concordance and health status) outcomes. Subjects ages 10-18 years are targeted for the HABIT intervention because transition of responsibility for self-management occurs *throughout this* time <sup>59,92,93</sup>. The PRECEDE portion of the PRECEDE-PROCEED Model of health program planning and evaluation <sup>38</sup> guides the qualitative interviews

and analysis of Aim 4. The model has been widely used in evaluation of health interventions such as physical activity<sup>94</sup> and obesity prevention.<sup>95,96</sup> In the proposed study, we use PRECEDE to gain better understanding of the effect of the HABIT intervention and its sustainability from the perspectives of the dyads who received the intervention and the CHWs who delivered it. These perspectives will provide context for interpretation of the quantitative findings and potential for broader dissemination of the HABIT intervention.

- **4. Setting.** Parent youth dyads will be recruited from 4 pediatric Sickle Cell Centers (Columbia University Medical Center, NY, NY; Montefiore Hospital, Bronx, NY; Cohen Children's Medical Center at Northwell Health, Queens, NY; Children's Hospital of Philadelphia, Philadelphia, PA). Each provides comprehensive multi-disciplinary care to youth with SCD. Considerable diversity in patient population exists within and among sites, including African American, African, West Indian and Latino families, as well as geographic and urban/rural location diversity. Pls at all participating sites have strong histories of successful recruiting and retaining of pediatric SCD patients for randomized trials, <sup>88,97-99</sup> despite potential barriers to trial enrollment. <sup>100-104</sup> While the volume of patients at each center varies (see **Resources**), we are confident that each site has sufficient youth who will both meet eligibility criteria and be interested in study participation (see **Enrollment Feasibility**) and will be successful in hiring experienced CHWs to deliver the intervention (see **C6**). While Cohen-Northwell has not worked directly with CHWs, they are experienced in working with the Sickle Cell-Thalassemia Patient Network, New York City's most established SCD patient group. Each site has wireless Internet in their clinic to allow use of iPad technology for direct entry of survey data into the HABIT RedCap database. All study visits will take place in the SCD outpatient clinic setting.
- **5. Study Participants.** To achieve **Aims 1-3**, a total of 104 youth-parent dyads meeting eligibility criteria (**Table 2**) will be recruited. Clinic rosters of youth ages 10-18 years and on HU therapy will be assessed for eligibility. Potentially eligible patients will be assessed for large decrease (≥20%) from Personal best HbF over the preceding 12 months. Those passing the initial screening will be telephoned for invitation to study participation. Of those interested, eligible dyads will be confirmed for full eligibility at their clinic visit. Those who meet all eligibility criteria will be offered enrollment until full enrollment is reached. Numbers and reasons for declining participation will be tracked at each site and cumulatively.

Table 2. Subject Eligibility and Exclusion Criteria

### **INCLUSION CRITERIA - YOUTH**

- 1. Sickle type HbSS or HbS-B<sup>0</sup> thalassemia
- 2. Age 10 through18 years (inclusive)
- 3. Currently prescribed HU ≥18 months (for identifying historical Personal best HbF)
- 4. Current HU dose is within 5% of dose at Personal Best HbF. For youth whose dose at Personal Best was ≥30mg/kg and whose current dose does not meet the 5% entry criterion, the dose of HU may be increased based on youth's current body weight not to exceed 30mg/kg. If subject meets all other entry criterion, subject may be recruited 3 months after dose adjustment
- Pre-enrollment HbF ≥15% below historical Personal best, based on mean of ≥2 HbF assessments over preceding 12 months
- 6. Youth able to speak/read English or Spanish

#### **INCLUSION CRITERIA - PARENT**

- 1. Parent/guardian speaks/reads English or Spanish
- 2. Parent/ legal guardian willing to participate
- 3. Family expects to reside in community for ≥ 1.5 years

### **EXCLUSION CRITERIA - YOUTH**

- 1. Youth not prescribed HU
- 2. <3 HbF assessments over past 12 months
- 3. Transfusion within 3 months preceding enrollment
- Final screen HbF (visit 0) of ≤15% decrease below Personal best HbF
- 5. Sexually active female ≥10 years and not using reliable contraception (due to HU teratogenic risk)
- 6. Pregnancy
- 7. Cognitive impairment (>2 levels below expected grade)
- 8. Youth not residing with parent/legal guardian
- 9. Sibling of a youth enrolled in this study

### **EXCLUSION CRITERIA – PARENT**

1. Parent/legal guardian does not reside with youth

For **Aim 4**, we will recruit two independent purposive samples of approximately 10 youth-parent dyads randomized to the HABIT intervention at each of 2 time points during their study experience: 6 months (perceived intervention impact) and 12 months (sustainability). The sample will represent dyads who make good progress to Personal Best HbF as well as those who continue to struggle with HU adherence.

### 6. Study Implementation Procedures

**Randomization.** A 1:1 randomization plan will be generated using computerized random number generator. A randomization plan will be generated for each site to achieve balanced randomization and will be maintained centrally at Columbia University Medical Center. Assignments to group will be placed in sequentially numbered

sealed envelopes stratified by site. Following subject consent and final screening, the site coordinator will contact Columbia PI for dyad assignment and study ID number.

### Recruitment and retention

**Subject enrollment.** Prior to study enrollment, parent/legal guardian consent and youth assent will be obtained by site coordinators for: study participation, release of pharmacy refill information for the year prior to study entry and for the duration of study participation, and (intervention arm only) for communication of HbF results and urgent clinical events to the CHW by study staff. A final screening will ensure that current HbF is consistent with levels over the past year. This screening will require the month 0 HbF level to be ≥15% below Personal best HbF (exclusion criterion 4). Randomization will await determination of this final eligibility criterion.

**Enrollment feasibility.** Full enrollment of 104 dyads (52 per study group) is expected based on excess number of eligible subjects (**Table 3**) and our HABIT enrollment experience during our feasibility trial. Three sites (CHOP, Cohen-Northwell and Montefiore) have capacity to enroll additional subjects in case of insufficient enrollment elsewhere. Despite compelling evidence of the value of HU therapy for youth with SCD, research has not translated into universal uptake. Table 3 provides detail regarding enrollment expectations from each site using data from our 2-site retrospective analysis to estimate the proportion of subjects who will meet the criterion of ±20% greater decrease from Personal best (i.e., 70%), and data from our feasibility trial to estimate the proportion of eligible children expected to consent (i.e., 58% of eligible subjects). With these sites we will achieve a sample size of 104 dyads, sufficiently powered to achieve the aims, while allowing for 20% subject attrition and/or receipt of blood transfusions (that alter HbF). Bi-monthly study visits is within the range of usual care frequency for patients on HU at each site.

Table 3. Estimation of target recruitment from each study site

| Table of Learnandi of tal got for almost from back orday one | | | | | |
|---|---|---|---|---|---|
| Site | # 10-18 yrs | # ≥20% below | # Estimated to | Target enrollment | CHW or related experience |
| | on HU | Personal best | consent | | |
| Columbia | 48 | 33 | 19 | 16 | HABIT study |
| Montefiore | 69 | 48 | 28 | 24 | HABIT study |
| Cohen-Northwell | 90 | 63 | 36 | 24 | No |
| CHOP | 200 | 140 | 81 | 40 | SCDAA |
| TOTAL | 461 | 322 | 186 | 104 | |

CHOP- Children's Hospital of Philadelphia; SCDAA –Sickle Cell Disease Association of America through their federally funded CHW program

**Retention** We expect high dyad retention based on low attrition (10.7%) during our HABIT feasibility trial; patients' long-term care at each SCD center; excellent enrollment and retention in previous SCD clinical trials under the PIs at each site; coordination of study visits with regular appointments; acceptability of text messaging for health interventions; and subject incentives weighted to study completion for extra time completing questionnaires (see Human Subjects). *Additionally, our planned 20% over-enrollment provides a cushion for subject attrition.* 

**Study Groups** Youth-parent dyads will be randomized to the HABIT intervention or the control group. They will be blinded to specific study hypotheses, even though they cannot be blinded to the assigned group. Both groups will have bi-monthly clinic visits over the 12 month study. In addition, intervention subjects will have visits with the CHWs as detailed below.

Data regarding laboratory assessment, hydroxyurea dosing and urgent hospital use will be collected at each visit by the study coordinator or his/her designee.

Control Group. Dyads

randomized to the control group will continue usual bi-monthly clinic-based care, including monitoring and review of HbF levels, and similar SCD team staff. They will receive the same educational materials (Appendix 5), complete the same questionnaires (Appendices 3, 4) and laboratory assessments as the Intervention group. They will



not receive CHW support or text messages.

**Intervention group.** The feasibility trial is now replicated in the proposed intervention trial (**Figure 2**) with the following additions: a) Dyad coaching on developing additional social support to enhance sustainability; b) More study sites (5 versus 2) and subjects (28 versus 104 dyads); and c) 6-month sustainability phase. CHW training and supervision are described below. The structured assessment for each CHW visit is found in Appendix 6.

Months 1-2: Month 1: One CHW visit at the home or other private location will initiate relationships between the CHW and youth-parent, individually and as a dyad to assess social, educational and self-management needs and identify barriers to HU adherence. CHWs will help dyads prioritize adherence barriers, address knowledge gaps about HU benefits/risks, and help dyads establish a shared plan for attaining HU adherence goals. Referrals for social services or other needs such as job training will be made to either the site's social services, community-based organization and/or other social service agencies in the community. Results of each bimonthly HbF testing months 0 through 8 and progress to personal best will be reviewed with the dyad by the CHW.

<u>Month 2</u>: CHW and dyad will jointly attend a SCD clinic visit to strengthen linkage with the SCD clinical service, and aid the dyad in reviewing plans to reduce adherence barriers. In addition, CHWs will meet with the dyad at home to focus on addressing adherence barriers, HU education and self-management strategies using a problem-solving approach. Additional service referrals will be made, as needed. Goals for youth self-management responsibility will be mutually agreed upon by the dyad, based on his/her age and capabilities, and regularly reviewed by the CHW.

<u>MONTHS 3-4</u>: CHWs will continue to support dyads on their roles and steps toward coordinated self-management, facilitate problem-solving to address barriers to a daily HU habit, and identify additional sources of personalized support for each dyad member (e.g. a relative or neighbor). Interim goals and progress toward goal achievement will be reviewed at each visit. Self-management issues will be addressed, depending on youth's age and developmental stage.

Month 3: The established CHW relationship will facilitate the CHW in coaching each dyad member to develop a text message reminder about taking HU: identify a daily cue-based habit to link to HU use, personalize text language, time of day and options of responses. Texts developed by dyads in the feasibility trial will serve as examples to help dyads develop a text message tailored to language, daily habit on which the cue is based and time of day preferences. CHW will clarify that messages are not their direct communication, but that they will receive timely information about texts from study staff. Contact with CHWs, if desired, can be made directly with CHWs via cell phone or text message.

Month 4: Begin daily text message reminders to parents and youth. Automated personalized text messages, delivered through MIR3 Notification solution, are intended to augment habit-forming behavior and extend ongoing support for a cue-based HU habit. The MIR3 system was used successfully during our HABIT feasibility trial and has been useful for Columbia faculty to automate communication with community-based research subjects 69,70,106,107.

Text messages will link HU reminders to the cue determined by each CHW-dyad, and will encourage a response such as "1" (taken) or "2" (not taken) or "3" (will take later), along with an option for sending free text, such as how they are feeling, problems with the medication, etc. Study staff will review text responses 2 times weekly and share them with the CHWs.

<u>Months 5-6</u>: Continued CHW focus on self-management, adherence and coaching to personal best HbF. Monthly CHW visits will continue. Using dyad text message response data from MIR3, weekly phone contact will be initiated in month 5 and continued through month 6 to provide positive reinforcement of HU adherence or to problem solve regarding why adherence has been a problem. To avoid habituation to text messages, the frequency of text messages will be negotiated based on preference of each dyad member at the end of month 5.

<u>MONTHS 7-12</u>: During the sustainability phase one CHW visit during month 9 will be scheduled to "boost" the effect of the intervention. This visit will be scheduled at the home or clinic, based on dyad preference. CHW focus will be limited to providing support by addressing questions or concerns that the dyad may have about issues related to adherence. During the sustainability phase, subjects will continue usual bi-monthly clinic visits, HbF and other laboratory assessment, and complete study questionnaires. We will track all dyad contact with the CHW during the sustainability phase.

Due to the COVID-19 pandemic and its implications for mental health distress, maladaptive behaviors (e.g. drinking, domestic violence), and food insecurity particularly in vulnerable populations, we will survey former and current parents and youth HABIT study participants using survey questions from the COVID-19 and mental health measurement working group at Johns Hopkins Bloomberg School of Public Health. All items are taken from valid survey instruments such as the CES-D (depression), GAD-7 (anxiety). We added 2 additional

items regarding food insecurity from the American Academy of Pediatrics recommended Hunger Vital Sign. The parent survey contains 18 items and the youth survey contains 15 items (an English and Spanish version of the parent and youth surveys are attached). Both surveys were translated to Spanish by our study team.

We propose to distribute the survey by either email or cell phone message that will provide a unique link to a REDCap survey. Using a script, the research coordinator at each site will contact both former and current study dyads of the HABIT Efficacy trial to describe the survey, participation is voluntary and that if a question makes them uncomfortable, they do not need to answer it. Current HABIT dyads will be contacted via telephone using a script; former HABIT dyads will be reconsented for participation by telephone using an information sheet. Participants will respond to the survey using their language of choice (English or Spanish). We propose to distribute the survey using the same platform, REDCap, as all other surveys administered as part of the HABIT study as soon as IRB approvals are obtained at each of the 4 study sites and again 2-4 months later to see the effect over time. Because of the sensitive nature of survey questions, research coordinator at each study site will monitor all survey responses as soon as possible and refer any "red flag" issues (e.g. domestic violence) to the social worker at the respective clinical site so that the patient may be referred for mental health services.

Qualitative Interviews with Dyad members. A purposive sample of parent-youth dyads from each clinical site will participate in individual interviews at 2 time points: after completing the 6-month study visit and at study completion (12 months). Interviews will be conducted by the coordinator at each site either face to face at the clinic or by telephone using uniform interview guides informed by the predisposing, enabling, and reinforcing constructs in Evaluate (PRECEDE) portion of the PRECEDE-PROCEED Model of health program planning and evaluation. Interviews for parents and youth will be conducted separately and each is expected to last approximately 20-30 minutes. Subjects will be compensated \$20 for their time. The interview guide for the 6 month interview will be directed to intervention impact. Interview guide questions for the 12 month interview will be geared toward the sustainability of the habit from the perspective of youth and parents. All interviews will be conducted in English, audiotaped, and transcribed for analysis. Based on clinic demographics at each site, most subjects will be fluent in English.

Sample questions will include:

- Tell me about the habit that you (your child) developed to make it easier to remember to take hydroxyurea every day? (reinforcing factor)
- What are some of the ways that you think your (your child's) health will improve through maintaining a hydroxyurea habit? (reinforcing factor)
- What do you perceive as barriers to maintaining a hydroxyurea habit? (predisposing factor); What are your ideas for how to maintain the habit that you (your child) have established? (enabling factor).

Focus groups with Community Health Workers: We will conduct 2 focus groups with all of the study CHWs at two time points: study mid-point (18 months) and end-point (36 months). Both focus groups will be conducted in English by webinar. CHWs will have become familiar with virtual meetings during monthly group supervision meetings as described below. Focus groups will be conducted in English, last approximately 60 minutes and will be led by Mr. Matos. The focus group interview guide questions will focus on the CHWs experiences with the dyads regarding the predisposing, enabling and reinforcing factors and their relationship to intervention impact and sustainability. Focus groups will be audiotaped and transcribed for analysis.

### **Intervention Training and Supervision**

**Training and Supervision.** A study orientation meeting of all site PIs and coordinators will be held at Columbia early in year 1 prior to subject enrollment. At that meeting, **Green** and **Smaldone** will present the study's main goals and strategies, including lessons learned from our feasibility trial, review the study protocol and address issues at any of the sites.

**CHW Training.** Two CHWs with prior CHW experience will be hired for the HABIT study at each site. The Co-PIs and site PIs will discuss leading candidates and will review the vetting process to ensure quality of CHWs and their prior training. Following hiring, CHWs from all sites will participate in a 4-day training session at Columbia led by **Matos**<sup>66</sup> (see LOS). Training will use the structured training curriculum from the HABIT feasibility study.<sup>31</sup> The first 2 days will serve as a "refresher" regarding CHW core concepts such as role and responsibility, engagement with families, and role boundaries. Days 3 and 4 of training will provide project-specific training, to include goals, rationale and approach by the HABIT study, schedule and goal of each CHW visit, information about SCD and HU (**Smaldone** and **Green** with **Matos**). Project specific skills, e.g., establishing relationships with dyads, helping dyads to work together to address barriers to HU and identify established daily patterns on which to build a HU habit, communication with the medical team will be

addressed through discussion and role playing. **Stennett** will discuss the importance of community support and resources for families faced with chronic illness (see LOS). **Bruzzese** will work with the group regarding motivational interviewing skills and self-management expectations for youth at varying age levels. The added benefit of group training is for the CHWs form a group allied for sharing experiences during supervision sessions over the course of the project. For any "red flag" issues (truancy, depression, drug use, potential violence), CHWs will be directed to immediately inform their site coordinator for referral to the clinic's social services.

**Supervision**. CHWs will have weekly ongoing supervision sessions to ensure high quality support to families, study fidelity, CHW progress with dyads and challenges to adherence, and detection of any barriers to progress towards an HU habit. Supervision schedule will include: a) bi-weekly site meetings with their coordinator to problem-solve for logistics of visits and the relationships with dyads, discuss on-going barriers to progress and reinforce the communication of HbF levels to dyads. b) Monthly site meetings jointly with their PI and coordinator will review additional study information and other social or medical issues; c) **Matos** (with **Smaldone** and **Green**) will lead monthly CHW group supervision sessions delivered via webinar for all CHWs to reinforce training components and ongoing case supervision; and d) At quarterly sessions, additional input to the CHWs on community-based intervention will be provided by **Stennett**. CHWs will share their experiences in delivering the intervention and will learn from the collective experiences.

If youth-parent dyads display unresolved conflict regarding self-management or other youth-parent relationship issues, **Matos** and **Bruzzese** will guide the approach of the staff and CHWs. Each site PI will meet with their respective CHWs a minimum of once per month with site coordinators the remaining weeks for CHW caseload updates, communicate with CHWs regarding subject HbF progress, information that may trigger clinical or social worker contact (e.g. turmoil in the home, missed school due to recurring disease symptoms or truancy), and to review all CHW visit forms and automated text messaging reports.

Treatment Fidelity will be assured through a structured intervention protocol (Figure 2 and Appendix 6), ongoing CHW supervision and monthly communication with site PIs and study coordinators. The HABIT operations manual contains: CHW encounter forms to structure and document the content of each scheduled encounter, monthly schedules and objectives to guide family discussion, key messages to promote HU adherence and youth-parent self-management partnership, exemplars of cues for text messaging reminders, and information for families on SCD and HU to be reviewed with dyads. CHW delivery of intervention and completed visit forms will be reviewed weekly during supervision. Feedback and guidance will be provided to CHWs for each dyad. Monthly conference calls will be held each for coordinators and for site PIs to oversee enrollment schedules, scheduling and logistics of home visits, obtaining pharmacy refill data, and study procedures and to problem-solving, as needed. To assure validity of HbF values, the subject's transfusion history will be reviewed during each coordinator call. Levels will be discarded if the subject had been transfused within the preceding 90 days, per standard HU protocols.

Variables and Operational Definitions: Table 4 overviews the variables including HbF levels and standard blood work for clinical monitoring, their relationship within the revised Self and Family Management

**Table 4. Study Measurement and Tools** 

| Concept/Variable | Р | Υ | Month | |
|---|---|---|---|---|
| Facilitators and Barriers | | | | |
| Health Status | | | | |
| Personal best HbF | Personal best HbF Highest historical HbF; Medical record | | • | 0 |
| Pre study HbF | Mean Preceding 12 month average of ≥3 HbF±standard deviation; Medical record | | • | 0 |
| Decrease from personal best | | | • | 0 |
| Past year's urgent medical | Hospitalization, ER visits, total hospital length of stay and | | • | 0 |
| service use | transfusions for past 12 months: Medical record | | | |
| Past year's HU adherence | Pharmacy refill (proportion of days covered) for past 12 months | | • | 0 |
| Health and HU monitoring | | | | |
| HbF | | | • | 0, 2, 4, 6, 9, 12 |
| CBC with reticulocyte count | Hb, MCV, platelet and absolute retic count, WBC, ANC | | • | 0, 2, 4, 6, 9, 12 |
| Liver and renal function tests | Total and indirect bilirubin, AST, ALT, creatinine, BUN | | • | 0, 6, 12 |
| Personal/Lifestyle | | | | |
| Age; Gender | Years; Male/female; Demographic survey | • | • | 0 |
| Race/ethnicity | African American; Hispanic; Demographic survey | • | • | 0 |
| Grade level (youth) | 1 through 12; Demographic survey | | • | 0 |
| Parental education | <high (hs);="" college;="" demographic="" etc.="" graduate;="" hs="" p="" school="" survey<=""></high> | • | | 0 |
| Barriers to HU use | 25-125; higher score = more barriers; Medication Barriers scale | • | • | 0, 6, 12 |

| Proximal Outcomes | | | | |
|---|---|---|---|---|
| Behaviors | | | | |
| Self-management responsibility | 1-50; higher score = greater responsibility; SCD Family Responsibility | • | • | 0, 2, 4, 6, 9, , 12 |
| Personal best HbF progress | HbF change; Medical record | | • | 0, 2, 4, 6, 9, 12 |
| Adherence | Progress to Personal best HbF (biomarker) | | • | 0, 2, 4, 6, 9, 12 |
| | Pharmacy refill (proportion of days covered) Pharmacy records | | • | 0, 2, 4, 6, 9, 12 |
| Symptoms | Pain interference | • | • | 0, 2, 4, 6, 9, 12 |
| | Pain intensity | • | • | 0, 2, 4, 6, 9, 12 |
| | Fatigue | • | • | 0, 2, 4, 6, 9, 12 |
| | Depressive symptoms | | • | 0. 6, 12 |
| | Emotional distress - Depression | • | | 0. 6, 12 |
| Distal Outcomes | | | | |
| <u>Family</u> | | | | |
| Parent productivity | | | | |
| Work related | 1-10; higher score = greater lost productivity; RUQ | • | | 0, 2, 4, 6, 9, 12 |
| Non work related | 1-10; higher score = greater lost productivity; RUQ | • | | 0, 2, 4, 6, 9, 12 |
| Individual/Family Outcomes | | | | |
| Quality of life | Generic 0-100; higher score = greater quality of life; <i>PedsQL generic core scale</i> | • | • | 0, 4, 9, 12 |
| | Disease specific 0-100; higher score = greater quality of life; PedsQL Sickle Cell Disease Module | • | • | 0, 4, 9, 12 |
| Self-management concordance | Self-management areas with consensus of responsibility; 0-10 with higher score=better communication; SCD Family Responsibility | • | • | 0, 2, 4, 6, 9, 12 |
| School attendance | Less missed school (days/past 2 months); RUQ | • | • | 0, 2, 4, 6, 9, 12 |
| Health Care Use | | | | |
| Emergency room | Number ER visits in past 2 months; RUQ; Medical record | • | | 0, 2, 4, 6, 9, 12 |
| Hospitalization | Hospitalizations in past 2 months; RUQ; Medical record | • | | 0, 2, 4, 6, 9, 12 |
| Hospital length of stay (LOS) | Total LOS in past 2 months; RUQ; Medical record | | | |
| Urgent visits | Urgent outpatient visits/past 2 months; RUQ; Medical | • | | 0, 2, 4, 6, 9, 12 |
| Subject satisfaction | | | | |
| Participant feedback | Evaluation survey | • | • | 12 |

Abbreviations: HbF = Hemoglobin F; HU = Hydroxyurea; P = Parent; Y = Youth; 0 = enrollment; 2 = 2 months; 4 = 4 months; 6 = 6 months; 9 = 9 months; 12 = 12 months; PedsQL = Pediatric Quality of Life; RUQ = Resource Use Questionnaire;

framework,<sup>91</sup> operational definitions, data sources and timing of data collection. All self-report instruments are found in Appendices 3 and 4. All measures piloted in the R21-funded feasibility study were valuable and will be used again. The exception is the Morisky scale of self-report medication adherence. This scale was found to be inconsistent with more objective biomarker and pharmacy refill. To address this, we have added 3 pediatric Patient Reported Outcomes Measurement Information System (PROMIS) measures (pain interference<sup>109</sup>, pain intensity and fatigue) to capture self-report of fatigue<sup>110</sup> and impact of pain from a youth and parent perspective<sup>111</sup>. PROMIS measures have been validated across multiple disease types for children<sup>112</sup>, have been validated in youth with SCD with scores responsive to hospitalization for sickle pain and subsequent recovery.<sup>87</sup> All survey data will be added directly into RedCap by the study participants with the exception of the demographic survey. Since that survey contains name, address and other identifying information, parent subjects will complete this survey via paper. The coordinator at each site will transcribe de-identified responses into RedCap. The paper survey will be stored in a locked cabinet in the PIs office together with the consent and assent.

**Demographic questionnaire**: 29 item questionnaire obtains youth-parent demographic information, medication profile and 12 month prior resource use.

**Medication Barriers scales**: 25 (parent) and 26 item (youth) 5 point Likert scales with established content, construct, and internal consistency<sup>17</sup>. Notably, the scale has established criterion validity with medication adherence<sup>17</sup>. Parent and adolescent scales were modified by adding 9 HU specific items<sup>19</sup>.

**Sickle cell Family Responsibility Scale**: 10 items; adapted from the Diabetes Family Responsibility Questionnaire (DFRQ)<sup>63</sup>; measures youth-parent perceptions of who takes responsibility for self-management tasks, division of responsibility<sup>65,113</sup>, dyadic agreement<sup>63,114</sup>; established internal consistency and concurrent validity (English, Spanish)<sup>115</sup>. DFRQ was adapted for use in asthma<sup>116</sup>, inflammatory bowel disease<sup>117</sup>, HIV<sup>59</sup>.

**Resource Use Questionnaire:** 11 items; adapted for SCD from the Resource Utilization Questionnaire for Type 1 diabetes (RUQ-T1DM)<sup>118</sup> with established content and criterion validity; uses a societal perspective.

**PedsQL Generic Core Scale:** 23 item 5 point Likert scale; 2 versions for youth (ages 8-12; 13-18 years) with parallel parent proxy version. High internal consistency for instrument ( $\alpha$ =0.91) and subscales ( $\alpha$ =0.81-0.89)<sup>119</sup> and has been validated in youth with SCD<sup>120-123</sup>; validated in Spanish.

**PedsQL Sickle Cell Disease Module:** 43 item 5 point Likert scale; 2 versions for youth (ages 8-12; 13-18 years) with parallel parent proxy version. High internal consistency for instrument ( $\alpha$ =0.95) and subscales ( $\alpha$ =0.69-90)<sup>89</sup>; validated in Spanish (see **Preliminary Studies C2**).

**Pain Interference – Short Form:** 8 item 5 point Likert scale; developed as part of the *PROMIS* initiative; *T*-score scale with mean = 50 and standard deviation = 10<sup>109</sup>; youth and parent proxy versions; available in Spanish.

**Pain Intensity** – 1 item visual analogue scale; scores range from 1-10; developed as part of the *PROMIS* initiative; examines perception of intensity of pain for the past 7 days; youth and parent proxy versions; available in Spanish.

**Fatigue – Short Form**: 10 item 5 point Likert scale; developed as part of the PROMIS initiative; T-score scale with mean = 50 and standard deviation =  $10^{110}$ ; youth and parent proxy versions; available in Spanish.

**Depressive symptoms (youth)**: 8 item 5 point Likert scale; developed as part of the PROMIS initiative; *T*-score scale with mean = 50 and standard deviation = 10, available in Spanish. Youth with depressive symptom T scores greater than 2 standard deviations above the mean will be referred for mental health counseling.

**Emotional distress – depression**: 4 item 5 point Likert scale; developed as part of the PROMIS initiative; *T*-score scale with mean = 50 and standard deviation = 10, available in Spanish. Parents with emotional distress T scores greater than 2 standard deviations above the mean will be referred for mental health conseling.

**Evaluation survey**: 26 item (for intervention group; 8 items for control group) investigator developed survey; 5 point Likert scale to assess impact on self-management, usefulness of materials, quality of CHW interaction, text messaging, cue-based medication reminders, outcomes, projected long-term study impact on disease self-management; 4 open ended items.

**COVID-19 survey**: 18 item (parent) and 15 item (youth) survey to measure mental health, maladaptive behaviors and food insecurity experienced by participant during the COVID-19 pandemic. All items taken from previously validated surveys.

### **D** Analytic Plan

**Power and sample size analysis:** We estimated the statistical power to compare score changes from the baseline to the follow-up times (for testing both improvement and sustainability) between the intervention and the control groups using the mixed model described below. All power analyses were based on the mixed model with 2-sided test and  $\alpha < 0.05$ . We assume that the outcome measure had a high correlation coefficient of 0.7 at different times and the clustering with each site was low with an intra-cluster coefficient (ICC) of 0.1. We also assume that this study will have 4 sites and each site has 16 to 40 subjects (total 104 subjects at the start of study). In each site, subjects will be 1 to 1 randomly assigned to the intervention and the control group with 20% attrition rate by the  $12^{th}$  month. For the DID analysis, we will have 83.2% power to detect a medium effect size of 0.6. We also estimated the statistical power to compare the trend of score changes from the baseline to the end of follow-up between the intervention and the control groups for outcomes that will be measured every 2 months from month 0 to month 12 visit. We will have 85.6% power to detect a small effect size of 0.25.

# Data analytic plan by Study Aim Aims 1-3:

**Aim 1**: Improve daily hydroxyurea (HU) adherence measured by two *primary outcomes*: biomarker (approach or exceed a historical Personal best HbF) and pharmacy refill (proportion of days covered). <u>Hypothesis 1</u>: Compared to the control group, dyads randomized to the intervention will improve medication adherence at 6 months, with sustained improvement at 12 months.

**Aim 2**: Improve quality of life and self-management responsibility measured by three secondary outcomes: generic and disease-specific QOL and parent/youth concordance regarding delegation of self-management responsibility. <u>Hypothesis 2</u>: Compared to the control group, dyads randomized to the intervention will report improved quality of life and self-management responsibility concordance at 6 months, with sustained improvement at 12 months.

**Aim 3**: Improve health status measured by two *secondary outcomes*: acute hospital use (12 month hospital length of stay, admissions and emergency room visits) and self-reported disease symptoms (fatigue, pain interference and intensity). *Hypothesis 3.1*: Compared to the control group, dyads randomized to the intervention group will demonstrate decreased acute hospital use at 6 months, with sustained improvement at 12 months. *Hypothesis 3.2*: Compared to the control group, dyads randomized to the intervention group will report decreased disease symptoms at 6 months, with sustained improvement at 12 months.

**COVID-19 survey** - Data will be analyzed using descriptive statistics. "Red flag" responses (e.g. domestic violence) will be referred to clinic social worker for management. Parent and youth responses will be compared.

Data analysis will be led by **Jia**. Analyses are based on intention to treat. All randomized subjects will be included in the analyses regardless of whether they adhered to the intervention protocol. Descriptive statistics will be used to profile outcome measures at each data collection point for the intervention and control groups. Distributions of all outcome variables will be made at the observational level instead of at the subject level. Medication adherence and quality of life assessments will be made at the 0, 6, and 12 month visit. Some outcomes (HbF, parent/youth concordance) will be assessed every 2 months from 0 to 12 month visit. We will compare hospital length of stay, emergency room visits, and hospitalizations during 3 time periods: 0-6 to the year prior, months 0-6, and months 7-12. The main analysis will be difference-in-difference (DID), comparison of changes in outcomes at 6 month from 0 month (improvement) and 12 month from 0 month (sustainability) between the intervention and the control group. We will use linear mixed model or generalized linear mixed model. Linear mixed models are used for most continuous outcomes (e.g. QOL score) and generalized linear mixed models are for categorical outcomes (e.g. whether or not a subject had an urgent outpatient visit with logit link function) or for outcomes with skewed distribution (e.g. length of stay with log link function). We will incorporate a site-specific random effect in the mixed models for controlling for clustering within each site. The mixed models are also used for outcomes that will be assessed every 2 months from 0 to 12 month visit to exam the difference in trend during the follow-up period. The mixed model is used to address the hierarchical data structure of multiple observations for each subject and multiple subjects in each family (i.e. youth-parent dyads) as well as for repeated measured data.

**Missing data**: Attrition or other missing data (survey or invalid HbF result due to recent transfusion) will be addressed by a plan to: (1) Apply a mixed model to include all subjects in the analysis; (2) Conduct a sensitivity analysis to estimate magnitude and direction of bias by imputing missing outcomes; and (3) Ask dyads who do not complete follow-up interviews about their reasons why and include such information in the model to correct the bias.

**Aim 4**: Qualitatively explore impact and sustainability of the intervention on developing a daily medication (HU) habit from the perspectives of the community health workers and youth-parent-dyads using focus group and individual interviews (*exploratory aim*).

Data analysis will be conducted by **Smaldone**<sup>124-126</sup> and **Findley**<sup>37</sup> both experienced in qualitative analysis. Each focus group and individual interview will be transcribed. The research team will ensure the credibility, confirmability, dependability and transferability of the qualitative data. To assure credibility we will conduct peer debriefing and triangulate findings across data sources (focus group, individual interview, survey data), use member checking, sharing of data interpretation with participants for accuracy. Triangulation of findings will enhance confirmability of findings. The research team will maintain an audit trail and maintain extensive field notes to facilitate transferability of findings. All transcripts and field notes will be analyzed using NVivo<sup>TM</sup> (QSR International, Victoria, Australia) software. Data will be sorted into categories by PRECEDE constructs: predisposing, enabling, and reinforcing to allow better understanding of the impact and sustainability potential of the HABIT intervention.

**E. Scientific Rigor**: Our interdisciplinary team has an outstanding track record of rigorous study design and implementation, including our prior feasibility trial. Several measures will be employed to generate valid and generalizable knowledge and to minimize bias. These include: 1) To avoid bias in study patient demographics, including sex, ethnicity and any additional medical conditions, offering study enrollment to sequential eligible patients at each site until the site sample is filled; 2) A 5-site study across differing study settings in three states assures greater diversity in subjects and circumstance and greater generalizability; 3) A careful central process for randomization of subjects within each site to help prevent bias in study arm assignment; 4) Use of objective data for assessing HU adherence, including determination of HbF when not affected by transfusion<sup>33</sup> and obtaining pre-study and 12 month study data on medication refills (**Aim 1**); 5) Self-reporting outcomes to augment staff report on acute hospital use, in case patients receive urgent care at other institutions during the 12-month study (**Aim 4**).<sup>76</sup>

### F. Study limitations and alternative strategies

**Sufficient enrollment:** Planned 20% over-enrollment and minimizing subject attrition will support full enrollment. In addition, three participating sites (Montefiore, CHOP and Cohen-Northwell) have excess capacity in case other sites cannot fully enroll.

**Investigator and subject blinding**: As CHWs have a major role in the intervention, blinding is not possible. Our procedure for allocation concealment minimizes potential bias regarding group assignment. Further, blinding will be maintained during the data analysis process.

Sample size insufficient to compare the effect of individual intervention components, CHWs and text messaging: Capture of dyad replies to text messages recorded by MIR3, as well as post-intervention focus groups, will provide qualitative information about any additive impact from text messaging.

**Peer support for parents and youth:** is not provided. Attending a peer support group would be difficult for this multi-ethnic sample, on top of busy families and working parents. Coaching youth and parent to develop identify individual support is intended to establish longer-term social support.

**If intervention impact is not sustainable at 12 months**: extended intensity of CHW support would require further testing. Post-intervention focus groups would identify subject recommendations for future trial design.

**G. Study Timeline** 

| Study Timeline* | Y1 | | | | Y2 | | | | Y3 | | | | Y4 | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Q1 | Q2 | Q3 | Q4 | Q1 | Q2 | Q3 | Q4 | Q1 | Q2 | Q3 | Q4 | Q1 | Q2 | Q3 | Q4 |
| IRB review and<br>Approval | • | • | | | | | | | | | | | | | | |
| Hiring and training<br>Coordinators | • | • | | | | | | | | | | | | | | |
| Hiring and training CHWs | | • | • | | | | | | | | | | | | | |
| Subject<br>Enrollment | | | • | • | • | • | • | • | • | • | • | • | | | | |
| 0-6 month<br>Intervention | | | | • | • | • | • | • | • | • | • | • | | | | |
| 7-12 month<br>Sustainability | | | | | | • | • | • | • | • | • | • | • | • | | |
| Qualitative interviews | | | | | | • | • | • | • | • | • | • | • | • | | |
| Data Analysis | | | | | | · | · | | | | | | | | • | • |
| Dissemination | | | | | | | | | | | | | | | • | • |

**H. Dissemination Plan**: will include multiple peer-reviewed publications and presentations at national meetings of experts represented by our multi-disciplinary team. We will continue to mutually co-inform the Sickle Cell Disease Association of America (SCDAA) regarding our respective multi-state CHW programs (LOS **Banks**) for program dissemination and shared efforts for enhancement and sustainability. Other partnerships will be developed to facilitate the adaptation of HABIT to other chronic pediatric conditions in underserved communities.

#### References

- 1. Hassell KL. Population estimates of sickle cell disease in the U.S. Am J Prev Med. 2010;38(4 Suppl):S512-21. doi: 10.1016/j.amepre.2009.12.022.
- 2. Brousseau DC, Panepinto JA, Nimmer M, Hoffmann RG. The number of people with sickle-cell disease in the United States: national and state estimates. Am J Hematol. 2010;85(1):77-8. doi: 10.1002/ajh.21570.
- 3. Brousseau DC, Owens PL, Mosso AL, Panepinto JA, Steiner CA. Acute care utilization and rehospitalizations for sickle cell disease. JAMA. 2010;303(13):1288-94. doi: 10.1001/jama.2010.378.
- 4. Raphael JL, Mei M, Mueller BU, Giordano T. High resource hospitalizations among children with vaso-occlusive crises in sickle cell disease. Pediatr Blood Cancer. 2012;58(4):584-90. doi: 10.1002/pbc.23181.
- 5. Lanzkron S, Carroll CP, Haywood C, Jr. Mortality rates and age at death from sickle cell disease: U.S., 1979-2005. Public health reports. 2013;128(2):110-6. PubMed Central PMCID: PMC3560868.
- 6. Hamideh D, Alvarez O. Sickle cell disease related mortality in the United States (1999-2009). Pediatr Blood Cancer. 2013;60(9):1482-6. doi: 10.1002/pbc.24557.
- 7. Yawn BP, Buchanan GR, Afenyi-Annan AN, Ballas SK, Hassell KL, James AH, Jordan L, Lanzkron SM, Lottenberg R, Savage WJ, Tanabe PJ, Ware RE, Murad MH, Goldsmith JC, Ortiz E, Fulwood R, Horton A, John-Sowah J. Management of sickle cell disease: summary of the 2014 evidence-based report by expert panel members. JAMA. 2014;312(10):1033-48. doi: 10.1001/jama.2014.10517.
- 8. McGann PT, Ware RE. Hydroxyurea for sickle cell anemia: what have we learned and what questions still remain? Curr Opin Hematol. 2011;18(3):158-65. doi: 10.1097/MOH.0b013e32834521dd. PubMed Central PMCID: PMCPMC3181131.
- 9. Ware RE. How I use hydroxyurea to treat young patients with sickle cell anemia. Blood. 2010;115(26):5300-11. doi: 10.1182/blood-2009-04-146852. PubMed Central PMCID: PMCPMC2902131.
- 10. Candrilli SD, O'Brien SH, Ware RE, Nahata MC, Seiber EE, Balkrishnan R. Hydroxyurea adherence and associated outcomes among Medicaid enrollees with sickle cell disease. Am J Hematol. 2011;86(3):273-7. doi: 10.1002/aih.21968.
- 11. Brandow AM, Panepinto JA. Monitoring toxicity, impact, and adherence of hydroxyurea in children with sickle cell disease. Am J Hematol. 2011;86(9):804-6. doi: 10.1002/ajh.22101. PubMed Central PMCID: PMC3804029.
- 12. Ritho J, Liu H, Hartzema AG, Lottenberg R. Hydroxyurea use in patients with sickle cell disease in a Medicaid population. Am J Hematol. 2011;86(10):888-90. doi: 10.1002/ajh.22134.
- 13. Thornburg CD, Calatroni A, Telen M, Kemper AR. Adherence to hydroxyurea therapy in children with sickle cell anemia. J Pediatr. 2010;156(3):415-9. doi: 10.1016/j.jpeds.2009.09.044. PubMed Central PMCID: PMC3901082.
- 14. Walsh KE, Cutrona SL, Kavanagh PL, Crosby LE, Malone C, Lobner K, Bundy DG. Medication adherence among pediatric patients with sickle cell disease: a systematic review. Pediatrics. 2014;134(6):1175-83. doi: 10.1542/peds.2014-0177. PubMed Central PMCID: PMC4243064.
- 15. Green NS, Manwani D, Qureshi M, Ireland K, Sinha A, Smaldone AM. Decreased fetal hemoglobin over time among youth with sickle cell disease on hydroxyurea is associated with higher urgent hospital use. Pediatr Blood Cancer. 2016. doi: 10.1002/pbc.26161.
- 16. Bogart LM, Wagner G, Galvan FH, Banks D. Conspiracy beliefs about HIV are related to antiretroviral treatment nonadherence among african american men with HIV. Journal of acquired immune deficiency syndromes. 2010;53(5):648-55. doi: 10.1097/QAI.0b013e3181c57dbc. PubMed Central PMCID: PMC2845717.
- 17. Simons LE, Blount RL. Identifying barriers to medication adherence in adolescent transplant recipients. Journal of pediatric psychology. 2007;32(7):831-44. doi: 10.1093/jpepsy/jsm030.
- 18. Tapp H, Hebert L, Dulin M. Comparative effectiveness of asthma interventions within a practice based research network. BMC health services research. 2011;11:188. doi: 10.1186/1472-6963-11-188. PubMed Central PMCID: PMC3176175.
- 19. Oyeku SO, Driscoll MC, Cohen HW, Trachtman R, Pashankar F, Mullen C, Giardina PJ, Velazco N, Racine AD, Green NS. Parental and other factors associated with hydroxyurea use for pediatric sickle cell disease. Pediatr Blood Cancer. 2013;60(4):653-8. doi: 10.1002/pbc.24381. PubMed Central PMCID: PMC3625668.
- 20. McQuaid EL, Everhart RS, Seifer R, Kopel SJ, Mitchell DK, Klein RB, Esteban CA, Fritz GK, Canino G. Medication adherence among Latino and non-Latino white children with asthma. Pediatrics. 2012;129(6):e1404-10. doi: 10.1542/peds.2011-1391. PubMed Central PMCID: PMC3362901.

- 21. Delgado EM, Cho CS, Gildengorin G, Leibovich SA, Morris CR. Parental asthma education and risks for nonadherence to pediatric asthma treatments. Pediatric emergency care. 2014;30(11):782-7. doi: 10.1097/PEC.000000000000259. PubMed Central PMCID: PMC4591748.
- 22. Wisk LE, Witt WP. Predictors of delayed or forgone needed health care for families with children. Pediatrics. 2012;130(6):1027-37. doi: 10.1542/peds.2012-0668. PubMed Central PMCID: PMC3507252.
- 23. Reach G. Role of habit in adherence to medical treatment. Diabet Med. 2005;22(4):415-20. doi: 10.1111/j.1464-5491.2004.01449.x.
- 24. McGrady ME, Hommel KA. Medication adherence and health care utilization in pediatric chronic illness: a systematic review. Pediatrics. 2013;132(4):730-40. doi: 10.1542/peds.2013-1451. PubMed Central PMCID: PMCPMC3784296.
- 25. Desai M, Oppenheimer JJ. Medication adherence in the asthmatic child and adolescent. Current allergy and asthma reports. 2011;11(6):454-64. doi: 10.1007/s11882-011-0227-2.
- 26. Taddeo D, Egedy M, Frappier JY. Adherence to treatment in adolescents. Paediatr Child Health. 2008;13(1):19-24. PubMed Central PMCID: PMCPMC2528818.
- 27. Salema NE, Elliott RA, Glazebrook C. A systematic review of adherence-enhancing interventions in adolescents taking long-term medicines. The Journal of adolescent health: official publication of the Society for Adolescent Medicine. 2011;49(5):455-66. doi: 10.1016/j.jadohealth.2011.02.010.
- 28. Quittner AL, Zhang J, Marynchenko M, Chopra PA, Signorovitch J, Yushkina Y, Riekert KA. Pulmonary medication adherence and health-care use in cystic fibrosis. Chest. 2014;146(1):142-51. doi: 10.1378/chest.13-1926.
- 29. Rothman RL, Mulvaney S, Elasy TA, VanderWoude A, Gebretsadik T, Shintani A, Potter A, Russell WE, Schlundt D. Self-management behaviors, racial disparities, and glycemic control among adolescents with type 2 diabetes. Pediatrics. 2008;121(4):e912-9. doi: 10.1542/peds.2007-1484.
- 30. Saha S, Jacobs EA, Moore RD, Beach MC. Trust in physicians and racial disparities in HIV care. AIDS patient care and STDs. 2010;24(7):415-20. doi: 10.1089/apc.2009.0288. PubMed Central PMCID: PMC3472674.
- 31. Smaldone A, Findley S, Bakken S, Matiz LA, Rosenthal SL, Jia H, Matos S, Manwani D, Green NS. Study protocol for a randomized controlled trial to assess the feasibility of an open label intervention to improve hydroxyurea adherence in youth with sickle cell disease. Contemporary clinical trials. 2016;49:134-42. doi: 10.1016/j.cct.2016.06.004.
- 32. Implementing NINR's Strategic Plan: Key Themes [cited 2016 Sept. 16]. Available from: https://www.ninr.nih.gov/aboutninr/keythemes .V-FtXbRbzpY.
- 33. Disparities: HealthyPeople.gov; [cited 2016 Sept. 20]. Available from: https://www.healthypeople.gov/2020/about/foundation-health-measures/Disparities.
- 34. Osterberg L, Blaschke T. Adherence to medication. N Engl J Med. 2005;353(5):487-97. doi: 10.1056/NEJMra050100.
- 35. Iuga AO, McGuire MJ. Adherence and health care costs. Risk management and healthcare policy. 2014;7:35-44. doi: 10.2147/RMHP.S19801. PubMed Central PMCID: PMC3934668.
- 36. Asche C, LaFleur J, Conner C. A review of diabetes treatment adherence and the association with clinical and economic outcomes. Clin Ther. 2011;33(1):74-109. doi: 10.1016/j.clinthera.2011.01.019.
- 37. Birmingham E, Catallozzi M, Findley SE, Vawdrey DK, Kukafka R, Stockwell MS. FluAlert: a qualitative evaluation of providers' desired characteristics and concerns regarding computerized influenza vaccination alerts. Preventive medicine. 2011;52(3-4):274-7. doi: 10.1016/j.ypmed.2011.01.008.
- 38. Gielen AC, McDonald EM, Gary TL, Bone LR. Using the PRECEDE/PROCEED Model to apply health behavior theories. In: Glanz K, Rimer BK, Viswanath K, editors. Health Behavior and Health Education: Theory, Research and Practice. 4th ed. San Francisco, CA: Jossey-Bass; 2008. p. 407-33.
- 39. Drotar D. Treatment adherence in patients with sickle cell anemia. J Pediatr. 2010;156(3):350-1. doi: 10.1016/j.jpeds.2009.10.035.
- 40. American Academy of P, American Academy of Family P, American College of P, Transitions Clinical Report Authoring G, Cooley WC, Sagerman PJ. Supporting the health care transition from adolescence to adulthood in the medical home. Pediatrics. 2011;128(1):182-200. doi: 10.1542/peds.2011-0969.
- 41. Walders N, Drotar D, Kercsmar C. The allocation of family responsibility for asthma management tasks in African-American adolescents. The Journal of asthma: official journal of the Association for the Care of Asthma. 2000;37(1):89-99.
- 42. DeBaun MR, Telfair J. Transition and sickle cell disease. Pediatrics. 2012;130(5):926-35. doi: 10.1542/peds.2011-3049.

- 43. Chaturvedi S, DeBaun MR. Evolution of sickle cell disease from a life-threatening disease of children to a chronic disease of adults: The last 40 years. Am J Hematol. 2016;91(1):5-14. doi: 10.1002/ajh.24235.
- 44. Steiner CA, Miller JL. Sickle Cell Disease Patients in U.S. Hospitals, 2004: Statistical Brief #21. Healthcare Cost and Utilization Project (HCUP) Statistical Briefs. Rockville (MD)2006.
- 45. Blood disorders and blood safety: HealthyPeople.gov; [cited 2016 Sept. 22]. Available from: https://www.healthypeople.gov/2020/topics-objectives/topic/blood-disorders-and-blood-safety/objectives.
- 46. Strouse JJ, Heeney MM. Hydroxyurea for the treatment of sickle cell disease: efficacy, barriers, toxicity, and management in children. Pediatr Blood Cancer. 2012;59(2):365-71. doi: 10.1002/pbc.24178. PubMed Central PMCID: PMCPMC3374046.
- 47. Brawley OW, Cornelius LJ, Edwards LR, Gamble VN, Green BL, Inturrisi C, James AH, Laraque D, Mendez M, Montoya CJ, Pollock BH, Robinson L, Scholnik AP, Schori M. National Institutes of Health Consensus Development Conference statement: hydroxyurea treatment for sickle cell disease. Ann Intern Med. 2008;148(12):932-8.
- 48. Darbari DS, Panepinto JA. What is the evidence that hydroxyurea improves health-related quality of life in patients with sickle cell disease? Hematology Am Soc Hematol Educ Program. 2012;2012:290-1. doi: 10.1182/asheducation-2012.1.290.
- 49. Fitzhugh CD, Hsieh MM, Allen D, Coles WA, Seamon C, Ring M, Zhao X, Minniti CP, Rodgers GP, Schechter AN, Tisdale JF, Taylor JGt. Hydroxyurea-Increased Fetal Hemoglobin Is Associated with Less Organ Damage and Longer Survival in Adults with Sickle Cell Anemia. PLoS One. 2015;10(11):e0141706. doi: 10.1371/journal.pone.0141706. PubMed Central PMCID: PMC4648496.
- 50. Smith WR, Ballas SK, McCarthy WF, Bauserman RL, Swerdlow PS, Steinberg MH, Waclawiw MA, Investigators of the Multicenter Study of Hydroxyurea in Sickle Cell A. The association between hydroxyurea treatment and pain intensity, analgesic use, and utilization in ambulatory sickle cell anemia patients. Pain medicine. 2011;12(5):697-705. doi: 10.1111/j.1526-4637.2011.01096.x.
- 51. Steinberg MH, McCarthy WF, Castro O, Ballas SK, Armstrong FD, Smith W, Ataga K, Swerdlow P, Kutlar A, DeCastro L, Waclawiw MA, Investigators of the Multicenter Study of Hydroxyurea in Sickle Cell A, Follow-Up MSHP. The risks and benefits of long-term use of hydroxyurea in sickle cell anemia: A 17.5 year follow-up. Am J Hematol. 2010;85(6):403-8. doi: 10.1002/ajh.21699. PubMed Central PMCID: PMC2879711.
- 52. Voskaridou E, Christoulas D, Bilalis A, Plata E, Varvagiannis K, Stamatopoulos G, Sinopoulou K, Balassopoulou A, Loukopoulos D, Terpos E. The effect of prolonged administration of hydroxyurea on morbidity and mortality in adult patients with sickle cell syndromes: results of a 17-year, single-center trial (LaSHS). Blood. 2010;115(12):2354-63. doi: 10.1182/blood-2009-05-221333.
- 53. Peretz PJ, Matiz LA, Findley S, Lizardo M, Evans D, McCord M. Community health workers as drivers of a successful community-based disease management initiative. Am J Public Health. 2012;102(8):1443-6. doi: 10.2105/AJPH.2011.300585. PubMed Central PMCID: PMCPMC3464827.
- 54. Uwemedimo OT, Arora G, Russ CM. New views on global child health: global solutions for care of vulnerable children in the United States. Curr Opin Pediatr. 2016;28(5):667-72. doi: 10.1097/MOP.0000000000000402.
- 55. Platt OS. Hydroxyurea for the treatment of sickle cell anemia. N Engl J Med. 2008;358(13):1362-9. doi: 10.1056/NEJMct0708272.
- 56. Zimmerman SA, Schultz WH, Davis JS, Pickens CV, Mortier NA, Howard TA, Ware RE. Sustained long-term hematologic efficacy of hydroxyurea at maximum tolerated dose in children with sickle cell disease. Blood. 2004;103(6):2039-45. doi: 10.1182/blood-2003-07-2475.
- 57. Hankins JS, Aygun B, Nottage K, Thornburg C, Smeltzer MP, Ware RE, Wang WC. From infancy to adolescence: fifteen years of continuous treatment with hydroxyurea in sickle cell anemia. Medicine (Baltimore). 2014;93(28):e215. doi: 10.1097/MD.000000000000215. PubMed Central PMCID: PMCPMC4603125.
- 58. Ferster A, Tahriri P, Vermylen C, Sturbois G, Corazza F, Fondu P, Devalck C, Dresse MF, Feremans W, Hunninck K, Toppet M, Philippet P, Van Geet C, Sariban E. Five years of experience with hydroxyurea in children and young adults with sickle cell disease. Blood. 2001;97(11):3628-32.
- 59. Naar-King S, Montepiedra G, Nichols S, Farley J, Garvie PA, Kammerer B, Malee K, Sirois PA, Storm D, Team PP. Allocation of family responsibility for illness management in pediatric HIV. Journal of pediatric psychology. 2009;34(2):187-94. doi: 10.1093/jpepsy/jsn065. PubMed Central PMCID: PMC2722122.
- 60. Anderson B, Ho J, Brackett J, Finkelstein D, Laffel L. Parental involvement in diabetes management tasks: relationships to blood glucose monitoring adherence and metabolic control in young adolescents with insulin-dependent diabetes mellitus. J Pediatr. 1997;130(2):257-65.

- 61. McQuaid EL, Kopel SJ, Klein RB, Fritz GK. Medication adherence in pediatric asthma: reasoning, responsibility, and behavior. Journal of pediatric psychology. 2003;28(5):323-33.
- 62. Orrell-Valente JK, Jarlsberg LG, Hill LG, Cabana MD. At what age do children start taking daily asthma medicines on their own? Pediatrics. 2008;122(6):e1186-92. doi: 10.1542/peds.2008-0292.
- 63. Anderson BJ, Auslander WF, Jung KC, Miller JP, Santiago JV. Assessing family sharing of diabetes responsibilities. Journal of pediatric psychology. 1990;15(4):477-92.
- 64. Treadwell MJ, Law AW, Sung J, Hackney-Stephens E, Quirolo K, Murray E, Glendenning GA, Vichinsky E. Barriers to adherence of deferoxamine usage in sickle cell disease. Pediatr Blood Cancer. 2005;44(5):500-7. doi: 10.1002/pbc.20290.
- 65. Anderson BJ, Brackett J, Ho J, Laffel LM. An office-based intervention to maintain parent-adolescent teamwork in diabetes management. Impact on parent involvement, family conflict, and subsequent glycemic control. Diabetes Care. 1999;22(5):713-21.
- 66. Findley SE, Matos S, Hicks AL, Campbell A, Moore A, Diaz D. Building a consensus on community health workers' scope of practice: lessons from New York. Am J Public Health. 2012;102(10):1981-7. doi: 10.2105/AJPH.2011.300566. PubMed Central PMCID: PMCPMC3490670.
- 67. Ayala GX, Vaz L, Earp JA, Elder JP, Cherrington A. Outcome effectiveness of the lay health advisor model among Latinos in the United States: an examination by role. Health Educ Res. 2010;25(5):815-40. doi: 10.1093/her/cvq035. PubMed Central PMCID: PMCPMC2948840.
- 68. Allen JK, Himmelfarb CR, Szanton SL, Bone L, Hill MN, Levine DM. COACH trial: a randomized controlled trial of nurse practitioner/community health worker cardiovascular disease risk reduction in urban community health centers: rationale and design. Contemporary clinical trials. 2011;32(3):403-11. doi: 10.1016/j.cct.2011.01.001. PubMed Central PMCID: PMCPMC3070050.
- 69. Stockwell MS, Kharbanda EO, Martinez RA, Vargas CY, Vawdrey DK, Camargo S. Effect of a text messaging intervention on influenza vaccination in an urban, low-income pediatric and adolescent population: a randomized controlled trial. JAMA. 2012;307(16):1702-8. doi: 10.1001/jama.2012.502.
- 70. Stockwell MS, Kharbanda EO, Martinez RA, Lara M, Vawdrey D, Natarajan K, Rickert VI. Text4Health: impact of text message reminder-recalls for pediatric and adolescent immunizations. Am J Public Health. 2012;102(2):e15-21. doi: 10.2105/AJPH.2011.300331. PubMed Central PMCID: PMCPMC3483980.
- 71. Estepp JH, Winter B, Johnson M, Smeltzer MP, Howard SC, Hankins JS. Improved hydroxyurea effect with the use of text messaging in children with sickle cell anemia. Pediatr Blood Cancer. 2014;61(11):2031-6. doi: 10.1002/pbc.25177.
- 72. Smaldone A, Stockwell MS, Osborne JC, Cortes Y, Bekele E, Green NS. Adolescent and parent use of new technologies for health communication: a study in an urban latino community. Journal of public health research. 2015;4(1):376. doi: 10.4081/jphr.2015.376. PubMed Central PMCID: PMC4407036.
- 73. Stockwell MS, Westhoff C, Kharbanda EO, Vargas CY, Camargo S, Vawdrey DK, Castano PM. Influenza vaccine text message reminders for urban, low-income pregnant women: a randomized controlled trial. Am J Public Health. 2014;104 Suppl 1:e7-12. doi: 10.2105/AJPH.2013.301620. PubMed Central PMCID: PMC4011110.
- 74. Gellad WF, Haas JS, Safran DG. Race/ethnicity and nonadherence to prescription medications among seniors: results of a national study. Journal of general internal medicine. 2007;22(11):1572-8. doi: 10.1007/s11606-007-0385-z. PubMed Central PMCID: PMC2219813.
- 75. Pai AL, Drotar D. Treatment adherence impact: the systematic assessment and quantification of the impact of treatment adherence on pediatric medical and psychological outcomes. Journal of pediatric psychology. 2010;35(4):383-93. doi: 10.1093/jpepsy/jsp073.
- 76. Anders DG, Tang F, Ledneva T, Caggana M, Green NS, Wang Y, Sturman LS. Hydroxyurea Use in Young Children With Sickle Cell Anemia in New York State. Am J Prev Med. 2016;51(1 Suppl 1):S31-8. doi: 10.1016/j.amepre.2016.01.001.
- 77. Hood KK, Rohan JM, Peterson CM, Drotar D. Interventions with adherence-promoting components in pediatric type 1 diabetes: meta-analysis of their impact on glycemic control. Diabetes Care. 2010;33(7):1658-64. doi: 10.2337/dc09-2268. PubMed Central PMCID: PMC2890378.
- 78. Kahana S, Drotar D, Frazier T. Meta-analysis of psychological interventions to promote adherence to treatment in pediatric chronic health conditions. Journal of pediatric psychology. 2008;33(6):590-611. doi: 10.1093/jpepsy/jsm128.
- 79. Creary SE, Gladwin MT, Byrne M, Hildesheim M, Krishnamurti L. A pilot study of electronic directly observed therapy to improve hydroxyurea adherence in pediatric patients with sickle-cell disease. Pediatr Blood Cancer. 2014;61(6):1068-73. doi: 10.1002/pbc.24931.

- 80. Inoue S, Kodjebacheva G, Scherrer T, Rice G, Grigorian M, Blankenship J, Onwuzurike N. Adherence to hydroxyurea medication by children with sickle cell disease (SCD) using an electronic device: a feasibility study. Int J Hematol. 2016;104(2):200-7. doi: 10.1007/s12185-016-2027-x.
- 81. Bruzzese JM, Kingston S, Sheares BJ, Cespedes A, Sadeghi H, Evans D. Feasibility and preliminary outcomes of a school-based intervention for inner-city, ethnic minority adolescents with undiagnosed asthma. Patient education and counseling. 2011;85(2):290-4. doi: 10.1016/j.pec.2010.09.019. PubMed Central PMCID: PMC3029508.
- 82. Bruzzese JM, Reigada LC, Lamm A, Wang J, Li M, Zandieh SO, Klein RG. Association of Youth and Caregiver Anxiety and Asthma Care Among Urban Young Adolescents. Acad Pediatr. 2016. doi: 10.1016/j.acap.2016.03.009.
- 83. Bruzzese JM, Sheares BJ, Vincent EJ, Du Y, Sadeghi H, Levison MJ, Mellins RB, Evans D. Effects of a school-based intervention for urban adolescents with asthma. A controlled trial. American journal of respiratory and critical care medicine. 2011;183(8):998-1006. doi: 10.1164/rccm.201003-0429OC. PubMed Central PMCID: PMC3086747.
- 84. Bruzzese JM, Unikel L, Gallagher R, Evans D, Colland V. Feasibility and impact of a school-based intervention for families of urban adolescents with asthma: results from a randomized pilot trial. Family process. 2008;47(1):95-113.
- 85. Stockwell MS, Hofstetter AM, DuRivage N, Barrett A, Fernandez N, Vargas CY, Camargo S. Text message reminders for second dose of influenza vaccine: a randomized controlled trial. Pediatrics. 2015;135(1):e83-91. doi: 10.1542/peds.2014-2475. PubMed Central PMCID: PMC4279072.
- 86. Dampier C, Barry V, Gross HE, Lui Y, Thornburg CD, DeWalt DA, Reeve BB. Initial Evaluation of the Pediatric PROMIS(R) Health Domains in Children and Adolescents With Sickle Cell Disease. Pediatr Blood Cancer. 2016;63(6):1031-7. doi: 10.1002/pbc.25944. PubMed Central PMCID: PMC4833539.
- 87. Dampier C, Jaeger B, Gross HE, Barry V, Edwards L, Lui Y, DeWalt DA, Reeve BB. Responsiveness of PROMIS(R) Pediatric Measures to Hospitalizations for Sickle Pain and Subsequent Recovery. Pediatr Blood Cancer. 2016;63(6):1038-45. doi: 10.1002/pbc.25931.
- 88. Wang W, Brugnara C, Snyder C, Wynn L, Rogers Z, Kalinyak K, Brown C, Qureshi A, Bigelow C, Neumayr L, Smith-Whitley K, Chui DH, Delahunty M, Woolson R, Steinberg M, Telen M, Kesler K. The effects of hydroxycarbamide and magnesium on haemoglobin SC disease: results of the multi-centre CHAMPS trial. Br J Haematol. 2011;152(6):771-6. doi: 10.1111/j.1365-2141.2010.08523.x.
- 89. Panepinto JA, Torres S, Bendo CB, McCavit TL, Dinu B, Sherman-Bien S, Bemrich-Stolz C, Varni JW. PedsQL sickle cell disease module: feasibility, reliability, and validity. Pediatr Blood Cancer. 2013;60(8):1338-44. doi: 10.1002/pbc.24491. PubMed Central PMCID: PMC4412167.
- 90. Grey M, Knafl K, McCorkle R. A framework for the study of self- and family management of chronic conditions. Nurs Outlook. 2006;54(5):278-86. doi: 10.1016/j.outlook.2006.06.004.
- 91. Grey M, Schulman-Green D, Knafl K, Reynolds NR. A revised Self- and Family Management Framework. Nurs Outlook. 2015;63(2):162-70. doi: 10.1016/j.outlook.2014.10.003.
- 92. Ingerski LM, Anderson BJ, Dolan LM, Hood KK. Blood glucose monitoring and glycemic control in adolescence: contribution of diabetes-specific responsibility and family conflict. The Journal of adolescent health: official publication of the Society for Adolescent Medicine. 2010;47(2):191-7. doi: 10.1016/j.jadohealth.2010.01.012. PubMed Central PMCID: PMCPMC2907244.
- 93. Helgeson VS, Reynolds KA, Siminerio L, Escobar O, Becker D. Parent and adolescent distribution of responsibility for diabetes self-care: links to health outcomes. Journal of pediatric psychology. 2008;33(5):497-508. doi: 10.1093/jpepsy/jsm081. PubMed Central PMCID: PMC3442285.
- 94. Slawta JN, DeNeui D. Be a Fit Kid: nutrition and physical activity for the fourth grade. Health Promot Pract. 2010;11(4):522-9. doi: 10.1177/1524839908328992.
- 95. Cole RE, Horacek T. Applying precede-proceed to develop an intuitive eating nondieting approach to weight management pilot program. J Nutr Educ Behav. 2009;41(2):120-6. doi: 10.1016/j.jneb.2008.03.006.
- 96. Manios Y, Grammatikaki E, Androutsos O, Chinapaw MJ, Gibson EL, Buijs G, Iotova V, Socha P, Annemans L, Wildgruber A, Mouratidou T, Yngve A, Duvinage K, de Bourdeaudhuij I, ToyBox-study g. A systematic approach for the development of a kindergarten-based intervention for the prevention of obesity in preschool age children: the ToyBox-study. Obesity reviews: an official journal of the International Association for the Study of Obesity. 2012;13 Suppl 1:3-12. doi: 10.1111/j.1467-789X.2011.00974.x.
- 97. Reid ME, El Beshlawy A, Inati A, Kutlar A, Abboud MR, Haynes J, Jr., Ward R, Sharon B, Taher AT, Smith W, Manwani D, Ghalie RG. A double-blind, placebo-controlled phase II study of the efficacy and safety

- of 2,2-dimethylbutyrate (HQK-1001), an oral fetal globin inducer, in sickle cell disease. Am J Hematol. 2014;89(7):709-13. doi: 10.1002/ajh.23725.
- 98. Ware RE, Davis BR, Schultz WH, Brown RC, Aygun B, Sarnaik S, Odame I, Fuh B, George A, Owen W, Luchtman-Jones L, Rogers ZR, Hilliard L, Gauger C, Piccone C, Lee MT, Kwiatkowski JL, Jackson S, Miller ST, Roberts C, Heeney MM, Kalfa TA, Nelson S, Imran H, Nottage K, Alvarez O, Rhodes M, Thompson AA, Rothman JA, Helton KJ, Roberts D, Coleman J, Bonner MJ, Kutlar A, Patel N, Wood J, Piller L, Wei P, Luden J, Mortier NA, Stuber SE, Luban NL, Cohen AR, Pressel S, Adams RJ. Hydroxycarbamide versus chronic transfusion for maintenance of transcranial doppler flow velocities in children with sickle cell anaemia-TCD With Transfusions Changing to Hydroxyurea (TWiTCH): a multicentre, open-label, phase 3, non-inferiority trial. Lancet. 2016;387(10019):661-70. doi: 10.1016/S0140-6736(15)01041-7.
- 99. Bajwa R, Schechter T, Soni S, Gassas A, Doyle J, Sisler I, Godder K, Tatman D, Rumelhart S, Domm J, Miao Y, Frangoul H. Outcome of children who experience disease relapse following allogeneic hematopoietic SCT for hematologic malignancies. Bone Marrow Transplant. 2013;48(5):661-5. doi: 10.1038/bmt.2012.209.
- 100. Haywood C, Jr., Bediako S, Lanzkron S, Diener-West M, Strouse J, Haythornthwaite J, Onojobi G, Beach MC, Investigators I. An unequal burden: poor patient-provider communication and sickle cell disease. Patient education and counseling. 2014;96(2):159-64. doi: 10.1016/j.pec.2014.05.013. PubMed Central PMCID: PMC4115582.
- 101. Haywood C, Jr., Diener-West M, Strouse J, Carroll CP, Bediako S, Lanzkron S, Haythornthwaite J, Onojobi G, Beach MC, Investigators I, Investigators I. Perceived discrimination in health care is associated with a greater burden of pain in sickle cell disease. Journal of pain and symptom management. 2014;48(5):934-43. doi: 10.1016/j.jpainsymman.2014.02.002. PubMed Central PMCID: PMC4198520.
- 102. Haywood C, Jr., Lanzkron S, Bediako S, Strouse JJ, Haythornthwaite J, Carroll CP, Diener-West M, Onojobi G, Beach MC, Investigators I. Perceived discrimination, patient trust, and adherence to medical recommendations among persons with sickle cell disease. Journal of general internal medicine. 2014;29(12):1657-62. doi: 10.1007/s11606-014-2986-7. PubMed Central PMCID: PMC4242876.
- 103. Haywood C, Jr., Lanzkron S, Diener-West M, Haythornthwaite J, Strouse JJ, Bediako S, Onojobi G, Beach MC, for the II. Attitudes toward clinical trials among patients with sickle cell disease. Clinical trials. 2014;11(3):275-83. doi: 10.1177/1740774513519876. PubMed Central PMCID: PMC4387103.
- 104. Stevens EM, Patterson CA, Li YB, Smith-Whitley K, Barakat LP. Mistrust of Pediatric Sickle Cell Disease Clinical Trials Research. Am J Prev Med. 2016;51(1 Suppl 1):S78-86. doi: 10.1016/j.amepre.2016.01.024. PubMed Central PMCID: PMC4916926.
- 105. Ware RE, Eggleston B, Redding-Lallinger R, Wang WC, Smith-Whitley K, Daeschner C, Gee B, Styles LA, Helms RW, Kinney TR, Ohene-Frempong K. Predictors of fetal hemoglobin response in children with sickle cell anemia receiving hydroxyurea therapy. Blood. 2002;99(1):10-4.
- 106. Kharbanda EO, Stockwell MS, Fox HW, Rickert VI. Text4Health: a qualitative evaluation of parental readiness for text message immunization reminders. Am J Public Health. 2009;99(12):2176-8. doi: 10.2105/AJPH.2009.161364. PubMed Central PMCID: PMCPMC2775765.
- 107. Kharbanda EO, Vargas CY, Castano PM, Lara M, Andres R, Stockwell MS. Exploring pregnant women's views on influenza vaccination and educational text messages. Preventive medicine. 2011;52(1):75-7. doi: 10.1016/j.ypmed.2010.10.009.
- 108. Tolan PH, Gorman-Smith D, Henry D, Schoeny M. The benefits of booster interventions: evidence from a family-focused prevention program. Prev Sci. 2009;10(4):287-97. doi: 10.1007/s11121-009-0139-8.
- 109. Varni JW, Stucky BD, Thissen D, Dewitt EM, Irwin DE, Lai JS, Yeatts K, Dewalt DA. PROMIS Pediatric Pain Interference Scale: an item response theory analysis of the pediatric pain item bank. The journal of pain: official journal of the American Pain Society. 2010;11(11):1109-19. doi: 10.1016/j.jpain.2010.02.005. PubMed Central PMCID: PMC3129595.
- 110. Lai JS, Stucky BD, Thissen D, Varni JW, DeWitt EM, Irwin DE, Yeatts KB, DeWalt DA. Development and psychometric properties of the PROMIS((R)) pediatric fatigue item banks. Quality of life research: an international journal of quality of life aspects of treatment, care and rehabilitation. 2013;22(9):2417-27. doi: 10.1007/s11136-013-0357-1. PubMed Central PMCID: PMC3695011.
- 111. Irwin DE, Gross HE, Stucky BD, Thissen D, DeWitt EM, Lai JS, Amtmann D, Khastou L, Varni JW, DeWalt DA. Development of six PROMIS pediatrics proxy-report item banks. Health and quality of life outcomes. 2012;10:22. doi: 10.1186/1477-7525-10-22. PubMed Central PMCID: PMC3312870.
- 112. DeWalt DA, Gross HE, Gipson DS, Selewski DT, DeWitt EM, Dampier CD, Hinds PS, Huang IC, Thissen D, Varni JW. PROMIS((R)) pediatric self-report scales distinguish subgroups of children within and

- across six common pediatric chronic health conditions. Quality of life research: an international journal of quality of life aspects of treatment, care and rehabilitation. 2015;24(9):2195-208. doi: 10.1007/s11136-015-0953-3. PubMed Central PMCID: PMC4531096.
- 113. Anderson BJ, Vangsness L, Connell A, Butler D, Goebel-Fabbri A, Laffel LM. Family conflict, adherence, and glycaemic control in youth with short duration Type 1 diabetes. Diabet Med. 2002;19(8):635-42.
- 114. Anderson BJ, Holmbeck G, Iannotti RJ, McKay SV, Lochrie A, Volkening LK, Laffel L. Dyadic measures of the parent-child relationship during the transition to adolescence and glycemic control in children with type 1 diabetes. Families, systems & health: the journal of collaborative family healthcare. 2009;27(2):141-52. doi: 10.1037/a0015759. PubMed Central PMCID: PMC2843423.
- 115. Hsin O, La Greca AM, Valenzuela J, Moine CT, Delamater A. Adherence and glycemic control among Hispanic youth with type 1 diabetes: role of family involvement and acculturation. Journal of pediatric psychology. 2010;35(2):156-66. doi: 10.1093/jpepsy/jsp045. PubMed Central PMCID: PMC2821010.
- 116. McQuaid EL, Penza-Clyve SM, Nassau JH, Fritz GK, Klein R, O'Connor S, Wamboldt F, Gavin F. The asthma responsibility questionnaire: Patterns of family responsibility for asthma management. Chilren's Health Care. 2010;30:183-99.
- 117. Greenley RN, Doughty A, Stephens M, Kugathasan S. Brief report: development of the inflammatory bowel disease family responsibility questionnaire. Journal of pediatric psychology. 2010;35(2):183-7. doi: 10.1093/jpepsy/jsp052.
- 118. Smaldone A, Tsimicalis A, Stone PW. Measuring resource utilization in patient-oriented comparative effectiveness research: a psychometric study of the Resource Utilization Questionnaire. Research and theory for nursing practice. 2011;25(2):80-106. PubMed Central PMCID: PMC3237636.
- 119. Varni JW, Seid M, Kurtin PS. PedsQL 4.0: reliability and validity of the Pediatric Quality of Life Inventory version 4.0 generic core scales in healthy and patient populations. Medical care. 2001;39(8):800-12.
- 120. Thornburg CD, Calatroni A, Panepinto JA. Differences in health-related quality of life in children with sickle cell disease receiving hydroxyurea. J Pediatr Hematol Oncol. 2011;33(4):251-4. doi: 10.1097/MPH.0b013e3182114c54. PubMed Central PMCID: PMCPMC3729442.
- 121. Dale JC, Cochran CJ, Roy L, Jernigan E, Buchanan GR. Health-related quality of life in children and adolescents with sickle cell disease. Journal of pediatric health care: official publication of National Association of Pediatric Nurse Associates & Practitioners. 2011;25(4):208-15. doi: 10.1016/j.pedhc.2009.12.006. PubMed Central PMCID: PMC3124665.
- 122. McClellan CB, Schatz J, Sanchez C, Roberts CW. Validity of the Pediatric Quality Of Life Inventory for youth with sickle cell disease. Journal of pediatric psychology. 2008;33(10):1153-62. doi: 10.1093/jpepsy/jsn036.
- 123. Panepinto JA, Pajewski NM, Foerster LM, Hoffmann RG. The performance of the PedsQL generic core scales in children with sickle cell disease. J Pediatr Hematol Oncol. 2008;30(9):666-73. doi: 10.1097/MPH.0b013e31817e4a44. PubMed Central PMCID: PMC2667700.
- 124. Poghosyan L, Nannini A, Smaldone A, Clarke S, O'Rourke NC, Rosato BG, Berkowitz B. Revisiting scope of practice facilitators and barriers for primary care nurse practitioners: a qualitative investigation. Policy, politics & nursing practice. 2013;14(1):6-15. doi: 10.1177/1527154413480889.
- 125. Ritholz MD, Smaldone A, Lee J, Castillo A, Wolpert H, Weinger K. Perceptions of psychosocial factors and the insulin pump. Diabetes Care. 2007;30(3):549-54. doi: 10.2337/dc06-1755.
- 126. Smaldone A, Ritholz MD. Perceptions of parenting children with type 1 diabetes diagnosed in early childhood. Journal of pediatric health care: official publication of National Association of Pediatric Nurse Associates & Practitioners. 2011;25(2):87-95. doi: 10.1016/j.pedhc.2009.09.003. PubMed Central PMCID: PMC3053084.